CLINICAL TRIAL: NCT00927342
Title: A Comparison of BioGlue and Vivostat in the Prevention of Air Leak in Thoracic Surgery
Brief Title: BioGlue or Vivostat in the Control of Air Leak in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Professor P Goldstraw, Department of Thoracic Surgery, Royal Brompton Hospital, London UK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2005LS001B
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-06

CONDITIONS: Thoracic Surgery; Air Leak
Keywords: Air leak; Thoracic Surgery; Sealants
MeSH Terms: interventions — Bio-glue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vivostat (Active Comparator)
  Interventions: Other: Vivostat
- BioGlue (Active Comparator)
  Interventions: Other: BioGlue

INTERVENTIONS:
Other: Vivostat — Patients with an air leak at the end of thoracic surgery despite conventional measures(diathermy, suturing and/or stapling) will receive Vivostat sealant applied to the surface of the lung in an attempt to eliminate air leak
  Arms: Vivostat
Other: BioGlue — Patients with an air leak at the end of thoracic surgery despite conventional measures(diathermy, suturing and/or stapling) will receive Bioglue sealant applied to the surface of the lung in an attempt to eliminate air leak
  Arms: BioGlue

SUMMARY:
Following lung surgery air may continue to leak from the surface of the lung. Chest drains are placed to allow this air to be removed safely and prevent the lung from collapsing. Drains need to remain until the air leak from the lung has ceased.

Air which continues to leak results in longer chest drainage times which cause increased discomfort and immobility for patients. These patients are at risk of secondary complications such as infection. Longer hospital stays and increased costs ensue. A randomised controlled trial (RCT) conducted at The Royal Brompton Hospital has shown clear benefits in the management of difficult air leak with the use of BioGlue. BioGlue is a surgical sealant applied to the surface of the lung at the time of surgery.

BioGlue is of bovine origin. Concerns exist regarding the potential risk of transmission of blood borne diseases with bovine derived medical products. Should a surgical adhesive without these potential risks prove as effective as BioGlue then its use could be commended.

The Vivostat System is a medical system that derives a sealant from the patient's own blood. A small study has shown that it may also be of benefit in the management of difficult air leaks. The principal aim of our RCT is to compare the duration of air leak, length of chest drainage and hospital stay associated with BioGlue to that of Vivostat.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and over)
* Males and females
* Patients undergoing any thoracic surgical procedure likely to result in alveolar air leak.
* Written informed consent

Exclusion Criteria:

* Age less than 18 years
* Pregnancy
* Breast feeding
* Previous treatment with BioGlue or Vivostat
* Inability to give informed consent
* Pneumonectomy
* Empyema
* Grade 0 air leak

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2005-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Duration of air leak | Days post-operatively
Duration of intercostal drainage | Days post-operatively
Duration of hospital stay | Days post-operatively

SECONDARY OUTCOMES:
Post-operative complications | Days and weeks following discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Thoracic Surgery, The Royal Brompton Hospital, London, United Kingdom